CLINICAL TRIAL: NCT02791932
Title: Exercise Intervention for Preventing Perinatal Depression
Brief Title: Effect of Exercise on Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R40MC29454
Record Dates: First submitted 2016-05-27; First posted 2016-06-07 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy; Postpartum Period; Depression
Keywords: Pregnancy; Postpartum period; Depression
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The intervention will last 8-10 months depending on when during pregnancy the participant is randomized. The intervention will consist of three components (i.e., telephone, print materials, and exercise log/goal setting) designed to increase exercise. Social Cognitive Theory (SCT) and Self-Determination Theory will guide the exercise intervention. The counseling sessions will be a collaboration between the counselor and participants on how to best integrate exercise into the participant's daily routine. Participants will receive 15 intervention phone calls lasting approximately 15-20 minutes each. There will be a one-month intensive phase (weekly contacts), followed by bi-weekly contacts for two months, and then monthly until delivery. Beginning at 6 weeks postpartum, bi-weekly contacts will resume through 3 months postpartum.
  Interventions: Behavioral: Exercise
- Usual Care (No Intervention): Participants in the usual care condition will follow their usual standard of care as suggested by their healthcare provider. Participants will complete the same assessments and incentives as the active interventions but will not receive the exercise counseling sessions. Following completion of the nine-month follow-up, the usual care arm can choose to receive a six-month version of the exercise intervention.

INTERVENTIONS:
Behavioral: Exercise — See description above.
  Arms: Exercise

SUMMARY:
Fifteen percent of women experience depression during pregnancy or postpartum (i.e., perinatal depression). Furthermore, 38% of low income women experience postpartum depression. Given few women with perinatal depression seek treatment, there is a need for innovative, low cost interventions that can be integrated within existing community-based programs serving women in need (e.g., low income women). The primary aim of this study is to examine the efficacy of a novel exercise intervention designed to prevent perinatal depression among women attending federally qualified health centers serving high risk women.

DETAILED DESCRIPTION:
Approximately 15% of women experience perinatal depression (depression during pregnancy or postpartum). Furthermore, 38% of low income women experience postpartum depression (Gree-Smith et al., 2012). Perinatal depression is associated with numerous maternal (e.g., weight retention), infant (e.g., poor infant-child bond), and lifespan (e.g., behavior problems) consequences (Barker et al., 2011, Herring et al., 2008, Hipwell et al., 2000). Psychosocial interventions are efficacious for perinatal depression; however, only 10% of women seek treatment (Oppo et al., 2009). There is a need for innovative, low cost interventions that can be integrated within existing community-based programs serving women in need (e.g., low income women). Preliminary evidence indicates that exercise may be a novel, efficacious intervention. The primary aim of this study is to examine the efficacy of a novel exercise intervention designed to prevent perinatal depression among women attending federally qualified health centers serving high risk women. Possible effects on gestational weight gain and retention will also be explored. This study will build upon the study team's previous work by recruiting low income women and integrating the intervention with community-based clinics. Participants (n=200) who are low income and pregnant (less than 20 weeks) will be randomly assigned to either a telephone-based intervention that has been previously shown to increase exercise among perinatal women (Lewis et al., 2011) or usual care.

With regard to the primary aim, the investigators predict that participants randomized to the exercise intervention will report fewer depressive symptoms (as measured by Edinburgh Postnatal Depression Scale) at 36 weeks gestation and three months postpartum than women in the usual care condition. The secondary aim is to examine the efficacy of an exercise intervention on moderating prenatal weight gain and facilitating postpartum weight loss. The investigators will also examine several potential mediators (e.g., depression coping, self-efficacy, perceived stress, sleep, fatigue) and the effect of the exercise intervention on maternal (e.g., hypertension, gestational diabetes, mode of delivery) and infant outcomes (e.g., birth weight, gestational age at delivery, breastfeeding, safe sleep).

ELIGIBILITY:
Inclusion Criteria:

* less than 20 weeks pregnant
* must speak English or Spanish
* willing to be randomly assigned to either of the two study arms
* healthcare provider consent
* access to a telephone (92% of low income women have access to a telephone and Minnesota offers free phone access for low income individuals; Fasts, 2015)
* being at risk for depression (defined as having a history of depression) but are not currently depressed.
* consistent with prior research, history of depression will be defined as ever being told by a healthcare provider that she has depression and/or being prescribed an antidepressant for depression.

Exclusion Criteria:

* less than 18 years of age
* currently exercising 60 or more minutes per week
* unable to exercise for 20 minutes continuously
* history of heart disease, lung disease, anemia, musculoskeletal problems (e.g., arthritis, gout, osteoporosis, or back, hip or knee pain that may interfere with exercising), poorly controlled hypertension, seizure disorder, exercise induced asthma, or any other medical condition that would make exercise unsafe
* taking medication that interferes with heart rate responses to exercise such as beta blockers; participating in another exercise or weight management study
* another member of the household participating in the study
* currently receiving antidepressant medication or psychotherapy for depression; - hospitalization for a psychiatric disorder during previous six months
* pregnant with multiple fetuses.
* participants depressed at the baseline assessment will be referred to their healthcare provider.
* there will have a safety protocol in place for worsening symptoms of depression and suicidal ideation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | Change from baseline to 3 months postpartum

SECONDARY OUTCOMES:
Postpartum Weight Retention | Change from baseline to 3 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Lewis, Minneapolis, Minnesota, United States